CLINICAL TRIAL: NCT05406336
Title: Machine Learning to Reduce Hypertension Treatment Clinical Inertia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K01HL151974 (NIH)
Record Dates: First submitted 2022-05-25; First posted 2022-06-06 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
Keywords: Uncontrolled blood pressure; Antihypertensive medication; Hypertension treatment; Clinical inertia; Machine learning
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No Information from Machine Learning Algorithm (No Intervention): The investigators will create case vignettes to assess clinician hypertension management behavior, specifically antihypertensive medication intensification among individuals with uncontrolled blood pressure (BP). This arm will not include information from a machine learning algorithm designed to predict uncontrolled BP at a follow up visit.
- Information from Machine Learning Algorithm (Experimental): The investigators will create case vignettes to assess clinician hypertension management behavior, specifically antihypertensive medication intensification among individuals with uncontrolled blood pressure (BP). This arm will include information from a machine learning algorithm designed to predict uncontrolled BP at a follow up visit about whether the algorithm predicts that the patient will have uncontrolled BP at the next visit.
  Interventions: Other: Predicted uncontrolled BP status (yes/no) at follow up visit, derived using a machine learning algorithm

INTERVENTIONS:
Other: Predicted uncontrolled BP status (yes/no) at follow up visit, derived using a machine learning algorithm — The investigators have created a machine learning algorithm to predict uncontrolled blood pressure (BP) status (yes/no) at a follow up visit among adults with uncontrolled BP at their current visit. The investigators will determine whether adding this information to a vignette describing a patient will increase the likelihood that a clinician will intensify antihypertensive medication treatment.
  Arms: Information from Machine Learning Algorithm

SUMMARY:
Among individuals with an uncontrolled BP at the current visit, the objective of this study is to compare clinical management of hypertension with and without information from a machine learning algorithm on whether a patient will have uncontrolled blood pressure at their next follow up visit through a case-vignette study.

DETAILED DESCRIPTION:
Among adults with uncontrolled blood pressure (BP) at a clinic visit, clinical inertia is common. Clinical inertia is defined as a failure of providers to initiate or intensify treatment (i.e., adding medication or increasing dosage) when guidelines indicate doing so. Prior studies report that clinicians intensify antihypertensive medication treatment in less than 20% of visits where intensification would have been clinically recommended. Thus, patients who have uncontrolled BP may not receive timely therapy to control their BP. To address this issue, the investigators will use a randomized design to test the hypothesis that clinicians will be more likely to intensify the hypertensive regimen and/or assess nonadherence for patients with uncontrolled BP at the current visit when presented with information that a patient is predicted to have uncontrolled BP at the next visit by a machine learning algorithm.

ELIGIBILITY:
Inclusion Criteria: practicing primary care clinicians who see patients (i.e., internal medicine, family medicine, attending physicians, nurse practitioners) will be eligible to participate -

Exclusion Criteria:

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Vignette #1 - antihypertensive medication treatment intensification | Immediately after clinical vignette
  A clinical vignette of a patient with uncontrolled blood pressure will be presented to clinicians. They will then be asked to assess wether they would intensify antihypertensive medication treatment. This will be assessed using a 5-point Likert scale with scores ranging from 1 ("Strongly disagree") to 5 ("Strongly agree"). Likert scale scores will be compared between clinicians in the control and intervention group.
Vignette #2 - antihypertensive medication treatment intensification | Immediately after clinical vignette
  A second clinical vignette of a patient with uncontrolled blood pressure will be presented to clinicians. They will then be asked to assess wether they would intensify antihypertensive medication treatment. This will be assessed using a 5-point Likert scale with scores ranging from 1 ("Strongly disagree") to 5 ("Strongly agree"). Likert scale scores will be compared between clinicians in the control and intervention group.
Vignette #3 - antihypertensive medication treatment intensification | Immediately after clinical vignette
  A third clinical vignette of a patient with uncontrolled blood pressure will be presented to clinicians. They will then be asked to assess wether they would intensify antihypertensive medication treatment. This will be assessed using a 5-point Likert scale with scores ranging from 1 ("Strongly disagree") to 5 ("Strongly agree"). Likert scale scores will be compared between clinicians in the control and intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Tajeu, DrPH, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No